CLINICAL TRIAL: NCT06986304
Title: Characterizing the Microvascular Environment of Bladder Cancer With Super-Resolution Ultrasound Localization Microscopy
Acronym: SR-ULM BC
Status: Not yet recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00117744
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The project will include 30 patients with bladder cancer who are candidates for bladder removal. After signing the consent form, the study team will collect some clinical data, such as age, past medical history, past surgical history, and information about your current disease.

At the day of surgery, after putting participants into sleep and before surgery begins, the study team will do a novel ultrasound called "Super-Resolution Ultrasound Localization Microscopy" to check if there is still disease in the bladder. The team will then compare the results of this investigational ultrasound with the final pathology and other imaging studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* Histological evidence of urothelial cancer of the bladder for which radical cystectomy is recommended as per the treating physician (e.g., MIBC or high-risk NMIBC, such as high-grade T1 BCG refractory and worrisome histological variants)

Exclusion Criteria:

* Known or suspected hypersensitivity to sulfur hexafluoride lipid microsphere or its components, such as polyethylene glycol (PEG).
* Pregnancy or breastfeeding
* Decline to participate in the study
* Participants who had serious allergic reactions to COVID-19 vaccination.
* Participants with unstable conditions such as hospital in-patients, ICU patients, or high-risk cardiac diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the clinic with bladder cancer for which a radical cystectomy is recommended.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Presence and stage of residual bladder cancer at the time of RC. | From enrollment to first post-cystectomy follow-up visit (1 month)
  The primary outcome variable is the presence and stage of residual bladder cancer at the time of RC. Statistical tests such as logistic regression will be applied to assess the accuracy of quantitative SR-ULM biomarkers in detecting residual bladder cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Abern, M.D., Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No